CLINICAL TRIAL: NCT05396339
Title: A Phase I/IIa Clinical Trial to Evaluate the Safety,Tolerability,Pharmacokinetics and Preliminary Effectiveness of IAE0972 in Patients With Advanced Malignant Solid Tumors.
Brief Title: A Clinical Trial to Evaluate the Effect of IAE0972 in Patients With Advanced Malignant Solid Tumors.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SUNHO（China）BioPharmaceutical CO., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IAE0972-I/IIa
Record Dates: First submitted 2022-05-19; First posted 2022-05-31 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Advanced Malignant Solid Tumor
Keywords: EGFR; IL10; Advanced Malignant Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase Ia - Dose escalation(Acceleration Stage) (Experimental): Phase Ia is an open, non-random, single-arm dose escalation design.
  Interventions: Drug: IAE0972
- Phase Ia - Dose escalation(3+3 Stage) (Experimental): Phase Ia is an open, non-random, single-arm dose escalation design.
  Interventions: Drug: IAE0972
- Phase Ib - Dose extension (Experimental): Phase Ib is an open, non-random, single-arm, multi-center research design.
  Interventions: Drug: IAE0972
- Phase IIa - Clinical Exploratory Stage (Experimental): The Phase IIa is planned to be divided into three indication groups, all of which are open, non-randomized, single-arm research design.
  Interventions: Drug: IAE0972

INTERVENTIONS:
Drug: IAE0972 — IAE0972 is an investigational product

SUMMARY:
This is a Phase I/IIa Clinical Trial to Evaluate the Safety,Tolerability,Pharmacokinetics and Preliminary Effectiveness of IAE0972 in Patients With Advanced Malignant Solid Tumors.

DETAILED DESCRIPTION:
The study includes three phases: dose escalation (Phase Ia), dose extension (Phase Ib), and clinical exploration (Phase IIa).First, the Phase Ia dose escalation will be carried out. After finishing the Phase 1a dose escalation, the Phase Ib dose extension study can be carried out in the MTD dose which is obtained from Phase 1a . After Phase Ia &1b are completed and RP2D is obtained, Phase IIa clinical exploratory research can be carried out.

ELIGIBILITY:
Inclusion Criteria:

* 1. Ability to provide informed consent and documentation of informed consent prior to initiation of any study-related tests or procedures that are not part of standard of care for the patient's disease. Patients must also be willing and able to comply with study procedures, including the acquisition of specified research specimens.

  2. Male or female, of any race, aged between 18 years and 80 years; 3. With histologically or cytologically confirmed locally advanced or metastatic solid malignant tumors, either refractory to standard therapy or for which no effective therapy was available.

  4. Measurable disease as determined by RECIST version 1.1 and documented by computed tomography (CT) and/or magnetic resonance imaging (MRI).

  5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. 6. Life expectancy ≥ 12 weeks. 7. Resolution of all chemotherapy or radiation-related toxicities to ≤ Grade 1 (with exception of ≤ Grade 2 alopecia, stable sensory neuropathy, or stable electrolyte disturbances that are managed by supplementation).

  8. Acceptable laboratory parameters as follows:
  1. Platelet count (PLT) ≥ 90 × 109/L without transfusion within 2 weeks prior to the initiation of investigational product.
  2. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L in the absence of any growth factor support within 2 weeks prior to the initiation of investigational product.
  3. International normalized ratio of prothrombin time (INR) ≤ 1.5 × upper limit of normal (ULN), activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.
  4. Hemoglobin (HGB) ≥ 90 g/L.
  5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 × ULN; for patients with hepatic metastases, ALT and AST ≤ 5.0 × ULN.
  6. Total bilirubin ≤ 1.5 × ULN, except patients with Gilbert's syndrome, who may enroll if the conjugated bilirubin is within normal limits.
  7. Serum creatinine < 1.5 × ULN, or estimated creatinine clearance ≥ 60 mL/min as measured or calculated using the Cockcroft-Gault formula.

     9. Female patients of childbearing potential (not surgically sterilized and between menarche and 1- year postmenopause) must have a negative serum or urine pregnancy test performed within 7 days prior to the initiation of investigational product administration. Further, female patients of childbearing potential must agree to use highly effective contraceptive measures (include hormonal contraceptives, intrauterine device or system, vasectomy, or tubal ligation) from the time of consent through 3 months after discontinuation of investigational product administration.

     10. Male patients with partners of childbearing potential must use barrier contraception. In addition, male patients should also have their partners use another method of contraception from the time of consent through 3 months after discontinuation of investigational product administration.

     Exclusion Criteria:
* 1. Known hypersensitivity (≥ Grade 3) to recombinant proteins or any excipient contained in the drug or vehicle formulation for IAE0972.

  2. History of another malignancy or a concurrent malignancy. Exceptions include patients who have been disease free for two years, or successfully treated for non-melanoma skin cancer, localized prostate cancer (Gleason Score < 6) or carcinoma in situ, for example cervical cancer in situ, are eligible.

  3. Treatment with any systemic anti-neoplastic therapy, radiation therapy or investigational therapy within 4 weeks prior to the initiation of investigational product administration, with the following exceptions:
  1. Nitrosourea or mitomycin C should be within 6 weeks prior to the initiation of investigational product administration.
  2. Oral fluoropyrimidines and small molecule targeted drugs should be within 2 weeks or 5 half-lives (whichever is later) prior to the initiation of investigational product administration.

     4. History of trauma or major surgery within 4 weeks prior to the initiation of investigational product administration.

     5. Treatment with corticosteroids (prednisone ≥ 10 mg per day or equivalent) or other immune suppressive drugs within the 14 days prior to the initiation of investigational product administration. Steroids for topical, ophthalmic, inhaled or nasal administration are allowed.

     6. Treatment with immunomodulatory agents, including but not limited to thymosin, interleukin-2 and interferon within 14 days prior to the initiation of investigational product administration.

     7. Vaccination with any live virus vaccine within 4 weeks prior to the initiation of investigational product administration.

     8. History of prior allogeneic bone marrow, stem-cell or solid organ transplantation.

     9. Active brain or leptomeningeal metastases. Patients with brain metastases are eligible if these have been treated and MRI or CT shows no evidence of progression for at least 8 weeks after treatment completion and within 4 weeks prior to the initiation of investigational product. Patients are not eligible if they required high doses of systemic corticosteroids that could result in immunosuppression (>10 mg/day prednisone equivalents) for at least 2 weeks prior to the initiation of investigational product.

     10. Evidence of active viral, bacterial, or systemic fungal infection requiring parenteral treatment within 7 days prior to the initiation of investigational product. Patients requiring any systemic antiviral, antifungal, or antibacterial therapy for active infection must have completed treatment no less than one week prior to the initiation of investigational product.

     11. Known history of hepatitis B or hepatitis C infection or known positive test for hepatitis B surface antigen, hepatitis B core antigen, or hepatitis C polymerase chain reaction (PCR).

     12. Known positive testing for human immunodeficiency virus (HIV) or history of acquired immune deficiency syndrome (AIDS).

     13. Clinically significant pulmonary compromise, including a requirement for supplemental oxygen use to maintain adequate oxygenation.

     14. History of clinically significant cardiovascular disease including but not limited to:

  <!-- -->

  1. Myocardial infarction or unstable angina within the 6 months prior to the initiation of investigational product.
  2. Stroke or transient ischemic attack within 6 months prior to the initiation of investigational product.
  3. Clinically significant cardiac arrhythmias, or a QTc prolongation to > 470 millisecond (ms) corrected by Fridericia's method based on a 12-lead electrocardiogram (ECG) in screening.
  4. Uncontrolled hypertension: systolic blood pressure (SBP) >180 mmHg, diastolic blood pressure (DBP) >100 mmHg.
  5. Congestive heart failure (New York Heart Association [NYHA] class III-IV).
  6. Pericarditis or clinically significant pericardial effusion.
  7. Myocarditis.
  8. Left ventricle ejection fraction (LVEF) < 50% by echocardiogram. 15. Any history of known or suspected autoimmune disease with the specific exceptions of vitiligo, resolved childhood atopic dermatitis, psoriasis not requiring systemic treatment (within the past 2 years), and patients with a history of autoimmune disease that are now clinically stable with replacement therapy and by laboratory testing.

     16. History of ≥ grade 3 immune-related adverse events (irAE) or Grade 2 immune-associated myocarditis accompanied with immunotherapy.

     17. Clinically uncontrolled effusion in the third space. 18. Known alcohol or drug dependence. 19. Dementia or altered mental status that would preclude understanding and rendering of informed consent.

     20. The female patient who is pregnant or breastfeeding, or expecting to conceive, AND the male patient who is expecting to father children within the projected duration of the trial, starting with the screening visit through 90 days after the last dose of trial treatment.

     21. Any issue that in the opinion of the investigator, would contraindicate the patient's participation in the study or confound the results of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06-24 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of IAE0972 in Phase I | 28 days after last medication, an average of 1 year
  MTD/R2PD ,Incidence and frequency of DTL; AE，SAE occurrence and frequency (according to NCI CTCAE 5.0)
Objective response rate (ORR) in Phase IIa | Baeline until disease progression, assessed up to 36 months
  To explore the effectiveness of IAE0972.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Cmax | after single dose , an average of 1 year
  PK parameters Cmax following single dose
Pharmacokinetic (PK) Css,max | after multiple doses , an average of 1 year
  PK parameters Css,max following multiple doses
Pharmacokinetic (PK) Css,min | after multiple doses , an average of 1 year
  PK parameters Css,min following multiple doses
Pharmacokinetic (PK) Css,av | after multiple doses , an average of 1 year
  PK parameters Css,av following multiple doses
Pharmacokinetic (PK) AUCss | after multiple doses , an average of 1 year
  PK parameters AUCss following multiple doses
Pharmacokinetic (PK) CLss | after multiple doses , an average of 1 year
  PK parameters CLss following multiple doses
Pharmacokinetic (PK) Vss | after multiple doses , an average of 1 year
  PK parameters Vss following multiple doses
Pharmacokinetic (PK) R | after multiple doses , an average of 1 year
  PK parameters R following multiple doses
Pharmacokinetic (PK) DF | after multiple doses , an average of 1 year
  PK parameters DF following multiple doses
Pharmacokinetic (PK) Cmin | after single dose , an average of 1 year
  PK parameters Cmin following single dose
Pharmacokinetic (PK) Tmax | after single dose , an average of 1 year
  PK parameters Tmax following single dose
Pharmacokinetic (PK) AUC0-t | after single dose , an average of 1 year
  PK parameters AUC0-t following single dose
Pharmacokinetic (PK) AUC0-∞ | after single dose , an average of 1 year
  PK parameters AUC0-∞ following single dose
Pharmacokinetic (PK) CL | after single dose , an average of 1 year
  PK parameters CL following single dose
Pharmacokinetic (PK) Vd | after single dose , an average of 1 year
  PK parameters Vd following single dose
Pharmacokinetic (PK) t1/2 | after single dose , an average of 1 year
  PK parameters t1/2 following single dose
Pharmacokinetic (PK) λz | after single dose , an average of 1 year
  PK parameters λz following single dose
Objective response rate (ORR) (Phase I ) | Baeline until disease progression or death, an average of 1 year
  To explore the preliminary effectiveness of IAE0972.
Overall survival (OS) (Phase I ) | Baeline until disease progression or death, an average of 1 year
  To explore the preliminary effectiveness of IAE0972.
Disease control rate (DCR) (Phase I ) | Baeline until disease progression or death, an average of 1 year
  To explore the preliminary effectiveness of IAE0972.
To evaluate the Immunogenicity of IAE0972 in patients with advanced malignant solid tumors (Phase I ) | Before each administration of dose cycle，an average of 1 year
  The frequency of anti-drug antibodies(ADA) against IAE0972
Progression-free survival（PFS) in Phase II | Baeline until disease progression or death,assessed up to 36 months
  To explore the effectiveness of IAE0972.
Overall survival (OS)in Phase II | Baeline until disease progression or death,assessed up to 36 months
  To explore the effectiveness of IAE0972.
Disease control rate (DCR) in Phase II | Baeline until disease progression or death,assessed up to 36 months
  To explore the effectiveness of IAE0972.
Immunogenicity of IAE0972 (Phase II ) | Before each administration of dose cycle,assessed up to 36 months
  The frequency of anti-drug antibodies(ADA) against IAE0972
Incidence of adverse event (AEs) and SAEs (Phase II) | After last medication,assessed up to 36 months
  To investigate the safety characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, M.D., Principal Investigator — Shanghai East Hospital; Yuping Sun, M.D., Principal Investigator — Affilated Cancer Hospital of Shandong First Medical University
Locations (2):
- China (2):
  - Affilated Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - Shanghai East Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No